CLINICAL TRIAL: NCT02866032
Title: A Multi-centre, Randomized, Two-armed, Parallel Group and Evaluator-blinded Study of Efficacy and Safety of Topical MOB015B in the Treatment of Mild to Moderate Distal Subungual Onychomycosis (DSO)
Brief Title: Study to Evaluate the Efficacy and Safety of Topical MOB015B in the Treatment of Mild to Moderate Distal Subungual Onychomycosis (DSO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: MOB015B-III
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Distal Subungual Onychomycosis
MeSH Terms: interventions — Ciclopirox

ARMS (2):
- MOB015B (Experimental)
  Interventions: Drug: MOB015B
- Ciclopirox 80 mg/g (Active Comparator)
  Interventions: Drug: Ciclopirox 80 mg/g

INTERVENTIONS:
Drug: MOB015B
  Arms: MOB015B
Drug: Ciclopirox 80 mg/g
  Arms: Ciclopirox 80 mg/g

SUMMARY:
The primary objective of this study is to evaluate the efficacy of topical MOB015B in patients with mild to moderate distal subungual onychomycosis (DSO).

The secondary objective is to evaluate the safety of topical MOB015B in patients with mild to moderate DSO.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 - 75 years of age
2. Distal subungual onychomycosis (DSO) of at least one of the great toenail(s) affecting 20% to 60% of the target nail
3. Positive culture for dermatophytes
4. Signed written informed consent

Exclusion Criteria:

1. Proximal subungual onychomycosis
2. Distal subungual onychomycosis of both great toenails where involvement has extended into the proximal portion of the target nail (unaffected proximal nail is less than 3 mm)
3. Target toenail thickness more than 3 mm
4. "Spike" of onychomycosis extending to eponychium of the target toenail
5. Presence of dermatophytoma (defined as thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the target nail
6. Other conditions than DSO known to cause abnormal nail appearance
7. Presence of toenail infection other than dermatophytes
8. Previous target toenail surgery with any residual disfigurement
9. Topical treatment of the nails with other antifungal medication or medical device within 6 weeks before screening/Visit 1
10. Systemic use of antifungal treatment within 6 months before screening/ Visit 1
11. Severe moccasin tinea pedis
12. Signs of severe peripheral circulatory insufficiency
13. Uncontrolled diabetes mellitus
14. Known immunodeficiency
15. Participation in another clinical trial with an investigational drug or device during the previous 3 months before Baseline/ Visit 2
16. Known allergy to any of the tested treatment products
17. A positive pregnancy test indicating pregnancy in a woman of childbearing potential at Baseline/ Visit 2
18. Females who are pregnant or breastfeeding
19. Pre-menopausal (last menstruation ≤ 1 year prior to screening) sexually active women who are of childbearing potential and are not practicing an acceptable method of birth control, or do not plan to continue practicing an acceptable method of birth control throughout the trial
20. Patients previously randomized in this study
21. History of, or current drug or alcohol abuse
22. Psychiatric condition that might limit the participation in the study and/or that lead to the assumption that the patient's ability to completely understand the consequences of consent is missing
23. Close affiliation with the investigator (e.g. a close relative) or persons working at a study site, or patient who is an employee of the sponsor's company
24. Patients who are institutionalized because of legal or regulatory order
25. Any diseases or circumstances in which the patient should not participate in the study in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2016-09; Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Complete cure of the target nail defined as negative fungal culture of dermatophytes, negative direct KOH microscopy and 0% clinical disease involvement at Week 52 | Week 52

CONTACTS AND LOCATIONS:
Locations (3):
- Multiple Locations, Germany
- Multiple Locations, Poland
- Multiple Locations, United Kingdom